CLINICAL TRIAL: NCT04211818
Title: Analysis of the Glycemic Profile of People Suffering From Compulsive Eating Disorders Aiming to Offer an Innovative Nutritional Approach
Brief Title: Analysis of the Glycemic Profile of People Suffering From Compulsive Eating Disorders Aiming to Offer an Innovative Nutritional Approach (GLUCOPULSE)
Acronym: GLUCOPULSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL18_0470
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2022-05

CONDITIONS: Bulimia; Binge Eating; Blood Glucose, Low; Crisis State; Compulsion
MeSH Terms: conditions — Bulimia; Compulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental)
  Interventions: Behavioral: Eating Behavior; Biological: Blood glucose records

INTERVENTIONS:
Behavioral: Eating Behavior — A dietary book will be given to the patient and will be filled by this one during 14 days
Biological: Blood glucose records — A glycemic sensor will be placed at the back of the patient's arm

SUMMARY:
Eating Disorders (ED) are a major public health problem. Current care remains only partially effective and the pathophysiology of the disorders remains to be deepened. With regard to compulsive ED (bulimia and binge eating disorder), our clinical experience suggests that one of the major triggers for crisis may be related to glycemia. In fact, bulimia could be considered as a vicious circle where the binge eating disorder is going to be followed by a food restriction in order to control weight , putting the subject in a situation of "energy deficiency" which will favor the emergence of new crises . Technological advances have resulted in the emergence of new measuring devices, such as "tracking", which records continuous glycemia, which would allow us to explore these clinical hypotheses.

DETAILED DESCRIPTION:
This is an open-label, exploratory, proof-of-concept study.

20 patients will be recruited from the day hospital of the Endocrinology and Nutrition Department of the University Hospital of Montpellier, Lapeyronie and from Emergencies and Post-psychiatric Emergencies Department.

During the inclusion visit, the dietician will explain to the patient the use of the dietary book and the glycemic sensor which will be allocated to it. The patient will also answer to self-questionnaires about his eating behavior.

No nutritional approach will be addressed so as not to alter the patient's eating behavior and not to influence the results.

They will be followed-up during 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Subject suffering from eating disorders with at least 3 episodes of bulimia per week for at least 2 months
* Subject affiliated to a health insurance or beneficiary of such a plan
* Subject able to understand the nature, purpose and methodology of the study
* Subject signed informed consent

Exclusion Criteria:

* Subject suffering from eating disorders such as anorexia nervosa
* Subject unable according to the investigator's opinion to keep updated a dietary book or to perform correctly the glycemic recordings
* Subject suffering from somatic pathology (ex: diabetes) or psychiatric pathology assessed by the MINI (ex : severe current major depressive episode) that may interfere with the protocol according to the the investigator
* Major subject legally protected (guardians or curators) or deprived of freedom by judicial or administrative order
* Pregnant or nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Frequency of episodes of bulimia (measured from the dietary book) according to the interstitial glucose levels | At the return of the dietary book (14 days after enrollment)
  Each information entered on the dietary book will be positioned on a chronological axis allowing to identify precisely when the eating disorder occurred

SECONDARY OUTCOMES:
Levels of impulse to make a crisis and food obsession and hunger depending on interstitial glucose levels | At the return of the dietary book (14 days after enrollment)
  Each information entered on the dietary book will be positioned on a chronological axis allowing to identify precisely when the eating disorder occurred
Dietary patterns | At enrollment
  Measured by the Emotional Appetite Questionnaire (EMAQ), 1 represent a food intake much smaller than usual ; 9 represent a food intake more significant than usual ; 5 represent a food intake as usual

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France